CLINICAL TRIAL: NCT01262365
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study of the Efficacy and Safety of Four 12-week Treatment Cycles (48 Weeks Total) of Epratuzumab in Systemic Lupus Erythematosus Subjects With Moderate to Severe Disease
Brief Title: Study of Epratuzumab Versus Placebo in Subjects With Moderate to Severe General Systemic Lupus Erythematosus
Acronym: EMBODY1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SL0009; 2010-018563-41 (EudraCT Number)
Record Dates: First submitted 2010-12-14; First posted 2010-12-17 (Estimated); Results first posted 2018-06-29 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Monoclonal antibody; B-Cell immunotherapy; Epratuzumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Weekly infusion) (Placebo Comparator): Placebo infusions delivered weekly for a total of 4 weeks over four 12-week treatment cycles
  Interventions: Drug: Placebo
- Epratuzumab 600 mg per week (Experimental): 600 mg infusions delivered weekly for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles
  Interventions: Drug: Epratuzumab
- Epratuzumab 1200 mg every other week (Experimental): 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles and placebo infusions delivered every other week for a total of 4 weeks over four 12-week treatment cycles
  Interventions: Drug: Epratuzumab; Drug: Placebo

INTERVENTIONS:
Drug: Epratuzumab — 600 mg infusions delivered weekly for a total of 4 weeks (cumulative dose 2400 mg) over four 12- week treatment cycles
  Arms: Epratuzumab 600 mg per week
Drug: Epratuzumab — 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles
  Arms: Epratuzumab 1200 mg every other week
Drug: Placebo — Placebo infusions delivered weekly for 4 weeks over four 12-week treatment cycles
  Arms: Epratuzumab 1200 mg every other week; Placebo (Weekly infusion)

SUMMARY:
The primary objective of the study is to confirm the clinical efficacy of epratuzumab in the treatment of subjects with Systemic Lupus Erythematosus (SLE)

ELIGIBILITY:
Inclusion Criteria:

* Positive antinuclear antibodies (ANA) at Screening (Visit 1)
* Current clinical diagnosis of Systemic Lupus Erythematosus (SLE) by American College of Rheumatology (ACR) criteria such that at least 4 of the 11 criteria are met
* Active moderate to severe SLE activity as demonstrated by the British Isles Lupus Assessment Group Index (BILAG)
* Active moderate to severe SLE disease as demonstrated by SLEDAI total score.
* On stable SLE treatment regimen, including mandatory corticosteroids and immunosuppressants or antimalarials

Exclusion Criteria:

* Subjects who are breastfeeding, pregnant, or plan to become pregnant
* Subjects with active, severe SLE disease activity which involves the renal system
* Subjects with active, severe, neuropsychiatric SLE, defined as any neuropsychiatric element scoring BILAG level A disease.
* Subjects with the evidence of an immunosuppressive state
* Subjects who, in the opinion of the investigator, are at a particularly high risk of significant infection
* History of malignant cancer, except the following treated cancers: cervical carcinoma in situ, basal cell carcinoma, or dermatological squamous cell carcinoma.
* Subjects receiving any live vaccination within the 8 weeks prior to screening (Visit 1).
* Subjects with history of infections, including but not limited to concurrent acute or chronic viral hepatitis B or C
* Subjects with substance abuse or dependence or other relevant concurrent medical condition
* Subjects with history of thromboembolic events within 1 year of screening Visit.
* Subjects with significant hematologic abnormalities
* Subject has received treatment with other anti- B cell antibodies within 12 months prior to screening (visit 1)
* Subject use of oral anticoagulant (not including) nonsteroidal anti-inflammatory drugs (NSAIDs) within 12 weeks prior to screening (Visit 1)
* Subject has previously participated in this study or has previously received epratuzumab treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2010-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCb Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (141):
- United States (50):
  - 069, Birmingham, Alabama
  - 063, Little Rock, Arkansas
  - 085, Escondido, California
  - 031, Los Angeles, California
  - 051, Los Angeles, California
  - 089, Los Angeles, California
  - 074, San Diego, California
  - 80, San Gabriel, California
  - 048, Aurora, Colorado
  - 037, Colorado Springs, Colorado
  - 039, Farmington, Connecticut
  - 042, Aventura, Florida
  - 090, Clearwater, Florida
  - 092, DeBary, Florida
  - 064, Jupiter, Florida
  - 082, Miami, Florida
  - 070, Ormond Beach, Florida
  - 084, Palm Harbor, Florida
  - 062, Tamarac, Florida
  - 050, Tampa, Florida
  - 087, Vero Beach, Florida
  - 044, Lawrenceville, Georgia
  - 052, Chicago, Illinois
  - 096, Indianapolis, Indiana
  - 060, Shreveport, Louisiana
  - 040, Baltimore, Maryland
  - 047, Saint Clair Shores, Michigan
  - 067, Las Cruces, New Mexico
  - 053, New York, New York
  - 077, Charlotte, North Carolina
  - 058, Durham, North Carolina
  - 061, Columbus, Ohio
  - 071, Middleburg Heights, Ohio
  - 041, Oklahoma City, Oklahoma
  - 076, Oklahoma City, Oklahoma
  - 097, Oklahoma City, Oklahoma
  - 032, Duncansville, Pennsylvania
  - 093, Philadelphia, Pennsylvania
  - 073, Pittsburgh, Pennsylvania
  - 094, Pittsburgh, Pennsylvania
  - 099, Charleston, South Carolina
  - 001, Columbia, South Carolina
  - 034, Simpsonville, South Carolina
  - 057, Memphis, Tennessee
  - 078, Austin, Texas
  - 098, Austin, Texas
  - 079, Dallas, Texas
  - 055, Houston, Texas
  - 036, Mesquite, Texas
  - 066, San Antonio, Texas
- Australia (5):
  - 426, Maroochydore, Queensland
  - 425, Malvern, Victoria
  - 429, Camperdown
  - 427, Clayton
  - 430, Liverpool
- Belgium (4):
  - 106, Brussels
  - 107, Brussels
  - 105, Leuven
  - 104, Liège
- Brazil (6):
  - 455, Campinas
  - 453, Porto Alegre
  - 451, Recife
  - 450, Rio de Janeiro
  - 452, Salvador
  - 454, São Paulo
- Bulgaria (6):
  - 201, Plovdiv
  - 200, Sofia
  - 202, Sofia
  - 203, Sofia
  - 204, Sofia
  - 205, Sofia
- Czechia (3):
  - 218, Olomouc
  - 216, Prague
  - 215, Zlín
- 226, Tallinn, Estonia
- France (4):
  - 113, Lille
  - 114, Nantes
  - 112, Paris
  - 116, Pessac
- Germany (5):
  - 127, Berlin
  - 128, Frankfurt
  - 126, Freiburg im Breisgau
  - 130, Hanover
  - 129, Plochingen
- India (3):
  - 351, Bangalore
  - 352, Hyderabad
  - 350, Lucknow
- Israel (9):
  - 378, Ashkelon
  - 376, Beersheba
  - 375, Haifa
  - 377, Haifa
  - 381, Jerusalem
  - 382, Kfar Saba
  - 380, Rehovot
  - 379, Tel Aviv
  - 383, Tel Litwinsky
- Italy (3):
  - 149, Ferrara
  - 148, Padua
  - 147, Torino
- Lithuania (2):
  - 155, Kaunas
  - 156, Klaipėda
- Mexico (4):
  - 475, Guadalajara
  - 476, Guadalajara
  - 478, Guadalajara
  - 480, Mérida
- Puerto Rico (2):
  - 091, Cidra
  - 086, San Juan
- Romania (5):
  - 263, Brasov
  - 260, Bucharest
  - 262, Bucharest
  - 264, Bucharest
  - 261, Cluj-Napoca
- Russia (3):
  - 285, Petrozavodsk
  - 284, Saint Petersburg
  - 281, Yekaterinburg
- South Korea (9):
  - 306, Busan
  - 303, Daegu
  - 309, Daegu
  - 308, Daejeon
  - 304, Incheon
  - 310, Jeonju
  - 301, Junggu
  - 307, Seoul
  - 302, Suwon
- Spain (8):
  - 165, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - 164, Bilbao, Vizcaya
  - 161, Barcelona
  - 162, Madrid
  - 163, Madrid
  - 166, Málaga
  - 177, Santander
  - 160, Seville
- Taiwan (5):
  - 325, Changhua
  - 326, Chiayi City
  - 328, Kaohsiung City
  - 329, Taichung
  - 330, Taipei
- United Kingdom (4):
  - 178, Brighton
  - 182, Doncaster
  - 179, Leeds
  - 181, Romford

REFERENCES:
- [Derived] Gottenberg JE, Dorner T, Bootsma H, Devauchelle-Pensec V, Bowman SJ, Mariette X, Bartz H, Oortgiesen M, Shock A, Koetse W, Galateanu C, Bongardt S, Wegener WA, Goldenberg DM, Meno-Tetang G, Kosutic G, Gordon C. Efficacy of Epratuzumab, an Anti-CD22 Monoclonal IgG Antibody, in Systemic Lupus Erythematosus Patients With Associated Sjogren's Syndrome: Post Hoc Analyses From the EMBODY Trials. Arthritis Rheumatol. 2018 May;70(5):763-773. doi: 10.1002/art.40425. Epub 2018 Apr 12. PMID 29381843
- [Derived] Clowse ME, Wallace DJ, Furie RA, Petri MA, Pike MC, Leszczynski P, Neuwelt CM, Hobbs K, Keiserman M, Duca L, Kalunian KC, Galateanu C, Bongardt S, Stach C, Beaudot C, Kilgallen B, Gordon C; EMBODY Investigator Group. Efficacy and Safety of Epratuzumab in Moderately to Severely Active Systemic Lupus Erythematosus: Results From Two Phase III Randomized, Double-Blind, Placebo-Controlled Trials. Arthritis Rheumatol. 2017 Feb;69(2):362-375. doi: 10.1002/art.39856. PMID 27598855

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in December 2010 and concluded in May 2015.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS).
Groups:
- Placebo (RS): Placebo infusions delivered weekly for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 1200 mg Every Other Week (RS): 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles and placebo infusions delivered every other week for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 600 mg Per Week (RS): 600 mg infusions delivered weekly for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles
Period: Overall Study
Arm/Group | Placebo (RS) | Epratuzumab 1200 mg Every Other Week (RS) | Epratuzumab 600 mg Per Week (RS)
Started | 266 | 262 | 265
Completed | 176 | 181 | 171
Not Completed | 90 | 81 | 94
Not completed — Lack of Efficacy | 35 | 30 | 47
Not completed — Protocol Violation | 3 | 1 | 1
Not completed — Lost to Follow-up | 3 | 7 | 6
Not completed — Withdrawal by Subject | 17 | 22 | 22
Not completed — Death | 1 | 2 | 1
Not completed — Adverse Event | 26 | 16 | 11
Not completed — sponsor decision | 1 | 1 | 0
Not completed — Randomization error | 1 | 0 | 2
Not completed — Non-compliance | 1 | 0 | 2
Not completed — Suspected pregnancy | 1 | 0 | 0
Not completed — Patient pregnant | 1 | 0 | 1
Not completed — Toxicity related to study drug | 0 | 1 | 0
Not completed — Cannot tolerate the protocol | 0 | 1 | 0
Not completed — Patient unavailable | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to the Safety Set.
Arm/Group | Placebo (Weekly Infusion) | Epratuzumab 1200 mg Every Other Week | Epratuzumab 600 mg Per Week | Total Title
Number analyzed (Participants) | 263 | 259 | 264 | 786
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 252 | 254 | 257 | 763
  >=65 years | 11 | 5 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.6) | 42.5 (11.8) | 42.3 (11.4) | 42.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 243 | 242 | 735
  Male | 13 | 16 | 22 | 51

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Subjects Meeting Treatment Response Criteria at Week 48 According to a Combined Response Index
Description: Percentages are based on the number of subjects in the relevant treatment group within the Full Analysis Set. The combined response index incorporated criteria for achievement of responder status from the: British Isles Lupus Assessment Group Index (BILAG-2004)- improvement from study entry or no worsening in other organ systems, Systemic Lupus Erythematosus Disease Activity Index (SLEDAI; Version 2000, also known as SLEDAI-2K) - no worsening compared to study entry, physician's global assessment of disease activity(PGA)- no worsening compared to study entry, and concomitant medications- no changes.
Time Frame: At Week 48
Population: The Full Analysis Set (FAS) consisted of all subjects in the Randomized Set (RS) who had received at least 1 partial dose of study drug, with the exception of 45 subjects who were randomized at Site 071, located in the USA, who were excluded from the FAS.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (Weekly Infusion) FAS: Placebo infusions delivered weekly for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 1200 mg Every Other Week (FAS): 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles and placebo infusions delivered every other week for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 600 mg Per Week (FAS): 600 mg infusions delivered weekly for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles
Arm/Group | Placebo (Weekly Infusion) FAS | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Per Week (FAS)
Number analyzed (Participants) | 249 | 244 | 248
percentage of participants | 34.1 | 39.8 | 37.5
Statistical Analysis 1: Comparison: Placebo (Weekly Infusion) FAS vs Epratuzumab 1200 mg Every Other Week (FAS); Odds Ratio: Epratuzumab/Placebo calculated using logistic regression with factors for treatment, region, and baseline disease status; Test type: Superiority; p = 0.175, Regression, Logistic; p-values have been calculated using logistic regression with factors for treatment, region, and baseline disease status; Odds Ratio (OR) = 1.307, 95% CI 2-sided [0.888 to 1.923]
Statistical Analysis 2: Comparison: Placebo (Weekly Infusion) FAS vs Epratuzumab 600 mg Per Week (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.442, Regression, Logistic; p-values have been calculated using logistic regression with factors for treatment, region, and baseline disease status; Odds Ratio (OR) = 1.164, 95% CI 2-sided [0.790 to 1.714]

2. Secondary Outcome: The Percent of Subjects Meeting Treatment Response Criteria at Week 24 According to a Combined Response Index
Description: as for outcome 1
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Weekly Infusion) FAS | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Per Week (FAS)
Number analyzed (Participants) | 249 | 244 | 248
percentage of participants | 33.7 | 43.0 | 39.1

3. Secondary Outcome: The Percent of Subjects Meeting Treatment Response Criteria at Week 12 According to a Combined Response Index
Description: as for outcome 1
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Weekly Infusion) FAS | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Per Week (FAS)
Number analyzed (Participants) | 249 | 244 | 248
percentage of participants | 31.3 | 42.2 | 39.9

4. Secondary Outcome: The Percent of Subjects Meeting Treatment Response Criteria at Week 36 According to a Combined Response Index
Description: as for outcome 1
Time Frame: At Week 36
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Weekly Infusion) FAS | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Per Week (FAS)
Number analyzed (Participants) | 249 | 244 | 248
percentage of participants | 33.3 | 41.8 | 35.1

5. Secondary Outcome: Change From Baseline in Daily Corticosteroid Dose at Week 24
Description: Subjects with a missing corticosteroid dose at any visit for any reason are counted in the Dose Increased or Missing Data category for that visit.
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Weekly Infusion) FAS | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Per Week (FAS)
Number analyzed (Participants) | 249 | 244 | 248
percentage of participants
  Dose decreased by >50% | 9.2 | 8.2 | 6.9
  Dose decreased >0% to <=50% | 10.8 | 16.4 | 14.9
  No change in dose | 52.2 | 50.0 | 50.8
  Dose increased or missing data | 27.7 | 25.4 | 27.4

6. Secondary Outcome: Change From Baseline in Daily Corticosteroid Dose at Week 48
Description: as for outcome 5
Time Frame: At Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Weekly Infusion) FAS | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Per Week (FAS)
Number analyzed (Participants) | 249 | 244 | 248
percentage of participants
  Dose decreased by >50% | 14.1 | 11.9 | 10.1
  Dose decreased >0% to <=50% | 10.4 | 14.3 | 12.5
  No chnage in dose | 38.6 | 37.7 | 37.9
  Dose increased or missing data | 36.9 | 36.1 | 39.5

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) were collected throughout the study (on or after first infusion of study drug and within 75 days of the last infusion), for an average of 4.4 years (starting in December 2010 and concluding in May 2015). The Safety Set (SS) will be utilized for TEAE reporting.
Description: The Safety Set consisted of all enrolled subjects who took at least 1 dose of study drug.
Arm/Group | Placebo (Weekly Infusion) | Epratuzumab 1200 mg Every Other Week | Epratuzumab 600 mg Per Week
All-Cause Mortality (participants affected / at risk) | 1/263 | 2/259 | 2/264
Serious Adverse Events (participants affected / at risk) | 48/263 | 44/259 | 45/264
Other Adverse Events (participants affected / at risk) | 144/263 | 153/259 | 141/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Weekly Infusion) (N=263) | Epratuzumab 1200 mg Every Other Week (N=259) | Epratuzumab 600 mg Per Week (N=264)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis lupus (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Bezoar (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 2 (2)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Serositis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (3) | 1 (1)
Lupus hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Myringitis bullous (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pyomyositis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 3 (3)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (3)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lupus encephalitis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mononeuropathy multiplex (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 2 (4) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Breast ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lupus vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Weekly Infusion) (N=263) | Epratuzumab 1200 mg Every Other Week (N=259) | Epratuzumab 600 mg Per Week (N=264)
Nausea (Gastrointestinal disorders) | 23 (28) | 30 (44) | 38 (49)
Diarrhoea (Gastrointestinal disorders) | 17 (19) | 21 (24) | 19 (28)
Fatigue (General disorders) | 10 (10) | 17 (20) | 12 (17)
Upper respiratory tract infection (Infections and infestations) | 30 (36) | 32 (38) | 32 (38)
Urinary tract infection (Infections and infestations) | 30 (41) | 25 (29) | 27 (41)
Nasopharyngitis (Infections and infestations) | 21 (26) | 20 (21) | 22 (29)
Sinusitis (Infections and infestations) | 13 (14) | 24 (24) | 15 (17)
Bronchitis (Infections and infestations) | 20 (23) | 12 (14) | 15 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (21) | 20 (28) | 14 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (14) | 19 (20) | 15 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (13) | 14 (18) | 9 (9)
Headache (Nervous system disorders) | 29 (38) | 34 (42) | 38 (58)
Dizziness (Nervous system disorders) | 11 (11) | 9 (10) | 16 (18)
Migraine (Nervous system disorders) | 3 (4) | 16 (19) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 13 (14) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 14 (16) | 8 (8)
Hypertension (Vascular disorders) | 11 (12) | 20 (21) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days